CLINICAL TRIAL: NCT03731923
Title: MR Value: Clinical Feasibility of Abbreviated MR Protocol for HCC Surveillance in High-risk Group
Brief Title: Abbreviated MRI for HCC Surveillance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Guerbet (Industry)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SNUH-2018-1426
Record Dates: First submitted 2018-11-04; First posted 2018-11-06 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Hepatocellular Carcinoma; Liver Cirrhosis; Chronic Hepatitis
Keywords: MRI; ultrasonography
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Cirrhosis; Hepatitis, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High risk group of HCC (Experimental): High risk group of HCC with chronic hepatitis or liver cirrhosis. Participants undergo biannual ultrasonography and annual abbreviated liver MRI.
  Interventions: Diagnostic Test: Biannual ultrasonography; Diagnostic Test: Annual abbreviated liver MRI

INTERVENTIONS:
Diagnostic Test: Biannual ultrasonography — Biannual liver ultrasonography for HCC surveillance, without contrast agent.
  Other Names: liver USG
Diagnostic Test: Annual abbreviated liver MRI — Abbreviated liver MRI using standard dose of extracellular contrast agent (Dotarem, Guerbet, France) on weight-based dosing. Table time targets 10 minutes.
  Other Names: Abbreviated liver MRI

SUMMARY:
This study aims to investigate the clinical feasibility of abbreviated liver MRI for HCC surveillance in a high-risk group.

ELIGIBILITY:
Inclusion Criteria:

* high risk of HCC development (chronic hepatitis B, chronic hepatitis C, liver cirrhosis)
* no history of HCC
* on surveillance of HCC using ultrasonography
* sign informed consent

Exclusion Criteria:

* history of HCC
* congestive hepatopathy
* iron deposition
* any absolute or relative contra-indication of contrast-enhanced MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity for detecting HCC | 12 months after last MRI
  Sensitivity for detecting HCC

SECONDARY OUTCOMES:
Table time of abbreviated MRI | 1 day after each MRI
  time from scan start and scan end
In-room time of abbreviated MRI | 1 day after each MRI
  interval between participants' walk-in and walk-out times
Specificity for detecting HCC | 12 months after last MRI
  Specificity for detecting HCC
Sensitivity for detecting early stage HCC | 12 months after last MRI
  Sensitivity for detecting early stage HCC (≤3cm, ≤3 tumors, or ≤5cm single tumor)
Specificity for detecting early stage HCC | 12 months after last MRI
  Specificity for detecting early stage HCC (≤3cm, ≤3 tumors, or ≤5cm single tumor)
Image quality of abbreviated liver MRI | 12 months after last MRI
  qualitative analysis on four-point scale

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No